CLINICAL TRIAL: NCT06099184
Title: A Phase 2, Multicenter, Prospective, Randomized, Double-Masked, Parallel Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), Compared to Aflibercept in Subjects With Diabetic Macular Edema (DME)
Brief Title: Study of EYP-1901 in Patients With Diabetic Macular Edema (DME)
Acronym: VERONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EYP-1901-202
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Macular Edema
Keywords: DME; EYP-1901; EyePoint
MeSH Terms: interventions — vorolanib; aflibercept

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EYP-1901 1343 µg (Experimental): EYP-1901 1343 µg, single dose
  Interventions: Drug: EYP-1901
- EYP-1901 2686 µg (Experimental): EYP-1901 2686 µg, single dose
  Interventions: Drug: EYP-1901
- Aflibercept (Active Comparator): Aflibercept 2 mg/0.05mL solution, single dose
  Interventions: Drug: Aflibercept 2Mg/0.05Ml Inj,Oph

INTERVENTIONS:
Drug: EYP-1901 — Intravitreal Injection
  Other Names: Vorolanib
  Arms: EYP-1901 1343 µg; EYP-1901 2686 µg
Drug: Aflibercept 2Mg/0.05Ml Inj,Oph — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
A prospective, randomized, single-masked study evaluating the ocular efficacy and safety of two doses of the EYP-1901 intravitreal insert compared to aflibercept

DETAILED DESCRIPTION:
A study to evaluate Efficacy and Safety of two doses of EYP-1901 in subjects with DME

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus in the study eye, with disease onset any time prior to the Screening Visit
* Previously treated with at least 1 intravitreal anti-VEGF in the last 6 months in the study eye at least 8 weeks prior to the Screening Visit.
* BCVA letter score of 35 letters (20/200 Snellen equivalent) to 75 letters (20/32 Snellen equivalent) in the study eye at the Screening Visit and at Baseline (Day 1).

Exclusion Criteria:

* Any current or history of ocular disease other than DME
* BCVA using ETDRS charts <30 letters (20/250 Snellen equivalent) in the fellow eye.
* Active ocular inflammation or active infection in either eye at Baseline (Day 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Time to first supplemental aflibercept injection following EYP-1901 dose at Baseline vs Aflibercept | Week 24
  Timing of supplemental injection

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) | Week 24
  Changes in BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Ribeiro, MD, Study Director — EyePoint Pharmaceuticals
Locations (6):
- United States (6):
  - EyePoint Investigative Site, Phoenix, Arizona
  - EyePoint Investigative Site, Lemont, Illinois
  - EyePoint Investigative Site, Hagerstown, Maryland
  - EyePoint Investigative Site, Reno, Nevada
  - EyePoint Investigative Site, Erie, Pennsylvania
  - EyePoint Investigative Site, Lynchburg, Virginia